CLINICAL TRIAL: NCT00065637
Title: PTH Once Weekly Research (POWR)
Brief Title: Once Weekly Parathyroid Hormone for Osteoporosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: N01 AR32268; N01AR002245-000 (NIH); NIAMS-092
Record Dates: First submitted 2003-07-29; First posted 2003-07-30 (Estimated); Last update posted 2013-02-05 (Estimated); Status verified 2013-02

CONDITIONS: Osteopenia; Osteoporosis
MeSH Terms: conditions — Bone Diseases, Metabolic; Osteoporosis | interventions — Teriparatide

ARMS (2):
- 1 (Experimental): Women will self-administer PTH injections daily for 4 weeks, then once weekly for 48 weeks
  Interventions: Drug: Teriparatide
- 2 (Placebo Comparator): Women will self-administer placebo injections daily for 4 weeks, then once weekly for 48 weeks
  Interventions: Drug: Placebo teriparatide

INTERVENTIONS:
Drug: Teriparatide — Synthetic human parathyroid hormone
  Arms: 1
Drug: Placebo teriparatide — Placebo injections
  Arms: 2

SUMMARY:
Daily parathyroid hormone (PTH) is approved by the FDA for the treatment of osteoporosis. This study will evaluate the safety and effectiveness of PTH when given once a week.

DETAILED DESCRIPTION:
In osteoporosis, skeletal bone mass and strength are so reduced that fractures occur after only modest levels of mechanical stress that would not harm normal bone. Fractures of the hip, spine, and wrists are most typical, though fractures of the ribs, pelvis, and humerus also occur. Research has shown that hip fractures cause a 10% to 20% increase in mortality, and the cost of all osteoporotic fractures is estimated to be $6.14 billion in health care costs and lost earnings per year. The most common form of osteoporosis is postmenopausal osteoporosis. A reduction in bone mineral density of approximately 1% to 2% per year is observed for the first 3 to 5 years after the onset of menopause, then 0.5% to 1% per year thereafter.

PTH was recently approved by the FDA as a daily treatment for osteoporosis. However, PTH must be self-injected, is very expensive, and has been associated with worrisome side effects. The currently approved formulation of daily PTH self-injections is practical for only a small proportion of people with osteoporosis. A once weekly formulation could significantly decrease cost, difficulty of administration, and risks and side effects associated with daily use of PTH. A once weekly injection by a caregiver would also make PTH accessible to populations for whom daily self-injection may not be practical, such as the very elderly or those in assisted living or nursing homes. This study will evaluate the safety and effectiveness of once weekly PTH dosing for women with osteoporosis.

Women will be randomized to receive either PTH or placebo. Women will self-administer injections daily for 4 weeks, then once weekly for 48 weeks. All women will receive calcium and vitamin D supplements daily. Women will visit the clinic six times over the course of a year and will provide urine and blood samples at each visit. Bone mineral density will be measured at 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Bone mineral density scan with a T-score between -1 and -2
* Willing to self-administer injections
* Postmenopausal

Exclusion Criteria:

* Medications to treat osteoporosis, including: hormone replacement therapy for more than one month in the 6 months prior to study, or for more than 12 months in the 2 years prior to study; alendronate, risedronate, or etidronate for more than 1 year anytime prior to study; calcitonin in the 3 months prior to study; taken raloxifene or tamoxifen in the last 6 months or for more than 1 year in the 2 years prior to study; fluoride for more than 1 month in the 5 years prior to study
* Bone fracture since menopause
* Femoral neck T-score below -2 AND lumbar spine T-score below -2.5 OR femoral neck T-score below -2.5 AND T-scores of both total hip and lumbar spine below -2

Ages: 45 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2003-12; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Bone mineral density | Months 6 and 12

CONTACTS AND LOCATIONS:
Overall Officials: Clifford Rosen, MD, Principal Investigator — Unity Health Toronto
Locations (1):
- St Joseph Hospital, Bangor, Maine, United States

REFERENCES:
- [Background] Brown SA, Rosen CJ. Osteoporosis. Med Clin North Am. 2003 Sep;87(5):1039-63. doi: 10.1016/s0025-7125(03)00065-8. PMID 14621330
- [Background] Rosen CJ. The cellular and clinical parameters of anabolic therapy for osteoporosis. Crit Rev Eukaryot Gene Expr. 2003;13(1):25-38. doi: 10.1615/critreveukaryotgeneexpr.v13.i1.30. PMID 12839095